CLINICAL TRIAL: NCT04935684
Title: Faecal Microbiota Transplantation for Prevention of Graft-versus-host Sisease After Allogeneic Stem Cell Transplantation for Haematological Malignancies
Brief Title: Faecal Microbiota Transplantation After Allogeneic Stem Cell Transplantation
Acronym: TMF-Allo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Ministry of Health, France (Other Government); French Society of Hematology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC N 2018 BAY; 2020-000673-24 (EudraCT Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-10

CONDITIONS: Acute Leukemia in Remission; Myelodysplastic Syndromes; Myeloproliferative Syndrome; Hodgkin Lymphoma; Lymphoma, Non-Hodgkin; Myeloma; Chronic Lymphocytic Leukemia
Keywords: Allogeneic hematopoietic stem cell transplantation; Hematologic malignancies; Graft versus Host Disease; Intestinal microbiota; Intestinal dysbiosis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Neoplasms, Plasma Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms; Graft vs Host Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: A group patients will receive Fecal Microbiota Transplantation (FMT) within 4 weeks following neutrophils recovery after the allogeneic hematopoietic stem cell transplantation procedure and a control group of patients will not receive FMT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Fecal Microbiota Transplantation (FMT) (Experimental): Patients randomized in the "FMT group" will received FMT. FMT product will be made by the the pharmacy of the Clermont-Ferrand University Hospital from stools of healthy volunteer donors within 6 hours after defecation in order to preserve the viability of the bacteria. The preparation will be standardized: 50g aliquots will be prepared and diluted in 250mL of 0.9% NaCl containing 10% glycerol, until a homogeneous suspension is obtained. The preparation will be rapidly frozen at -80°C until use, with a maximum shelf life of 18 months.
  Interventions: Drug: Fecal Microbiota Transplantation
- Group 2: no intervention (No Intervention): The comparator group will be constituted by patients randomized in the "no FMT" group. For ethical reasons, these patients will not receive any FMT and therefore no enema or colic preparation. No placebo will be administered. Prophylactic anti-infective treatments can be introduced at any time.

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Patients randomized in the "FMT group" will received FMT within 4 weeks following neutrophils recovery after the allo-HSCT procedure. The stool transplant will be done by enema. The day before FMT, patient will undergo bowel cleansing by ingestion of two liters of polyethylene glycol solution. The day of FMT, a colon cleanse enema will be performed in the morning and FMT will be delivered around two hours after the cleanse enema. This colic preparation is essential to optimize the results of FMT.
  The enema (50g of stools diluted in 250mL of NaCl 0.9%) will be performed by a qualified member of the study team (nurse) by using a rectal cannula (within 6 hours of thawing). The enema will have to be kept by the patient for as long as possible and at least 30 minutes.
  Arms: Group 1: Fecal Microbiota Transplantation (FMT)

SUMMARY:
The aim of this study is to assess the Fecal Microbiota Transplantation (FMT) efficacy in the prevention of allogeneic hematopoietic stem cell transplantation (allo-HSCT) complications and particularly Graft versus Host Disease (GvHD).

The hypothesis of this study is that allogeneic FMT may improve outcomes of these patients.

DETAILED DESCRIPTION:
The TMF-Allo study is a prospective, open-label, multi-center, parallel, randomized phase II clinical trial comparing a group patients with FMT and a control group of patients without FMT.

The main objective of this study is to assess the effect of allogeneic FMT versus no treatment on Graft-versus-host disease and Relapse-Free Survival (GRFS) at one year in adult patients treating with myelo-ablative allo-HSCT for haematologic malignancy.

The secondary objectives are to evaluate :

* Overall survival, progression-free survival at 1 and 2 years,
* The haematological evolution,
* The evolution of infections,
* The tolerance and safety of the TMF carried out in post-transplant,
* The evolution of the composition and diversity of the microbiota in allograft patients receiving TMF or not.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Men and women
* Patients affiliated with a social-security organization
* Patients undergoing a myelo-ablative allo-HSCT for a controlled haematologic malignant disease, with peripheral stem cells, whatever the type of donor (except cord blood)
* Signed and dated informed consent

Exclusion Criteria:

* Status of tumor progression at the time of allo-HSCT
* Inability to understand the protocol (linguistic barrier, cognitive difficulties)
* Medical history of another progressive cancer or occurrence in the 3 previous years (excluding basal cell carcinoma)
* Presence of a simultaneous serious and uncontrolled disease (severe cardiac, renal, hepatic or respiratory failure, severe sepsis)
* Fecal incontinence
* Participation in another clinical trial studying an allograft procedure including the type of graft, the type of immunosuppression, a preventive or a curative treatment of GvHD, or studying the effectiveness of a FMT in another indication.
* Pregnant women
* Patient under guardianship, curatorship or protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Graft-versus-host disease and Relapse-Free Survival (GRFS) rate after allogeneic hematopoietic stem cell transplantation | at Day 360 after allogeneic hematopoietic stem cell transplantation
  GRFS is a composite endpoint of GvHD-free/relapse-free survival in which events include grade II-IV acute GvHD, moderate and severe chronic GvHD, relapse, or death in the first year post-HSCT. GRFS will be measured at one year after allo-HSCT and compared between both groups of patients.

SECONDARY OUTCOMES:
Overall survival | At Day 360 and Day 720 after allogeneic hematopoietic stem cell transplantation
  Overall survival is defined as the time period between the date of randomization and the date of death, regardless of its cause.
Progression-free survival | At Day 360 and Day 720 after allogeneic hematopoietic stem cell transplantation
  Progression-free survival is defined as the time period between the date of randomization and the date of disease relapse or progression or death, regardless of its cause.
Haematopoietic reconstitution | At the time of haematopoietic reconstitution
  Haematopoietic reconstitution is assessed by: 1/ turnaround time of polynuclear neutrophils >0.5.10^9/L (first day within a period of three consecutive days); 2/ spontaneous platelet turnaround time >20.10^9/L (two days with no platelet transfusion within the previous three days); 3/ spontaneous platelet turnaround time >50.10^9/L (two days with no platelet transfusion within the previous three days); 4/ the number of transfusions of red blood cells and platelets between D0 and D100
Engraftment rates | At Day 30, Day 60, Day 90, Day 180, Day 360 and Day 720 after allogeneic hematopoietic stem cell transplantationday
  Engraftment rates are evaluated by a chimerism measure (by molecular biology)
Cumulative incidence of acute GvHD | At Day 360 after allogeneic hematopoietic stem cell transplantation
  Acute GvHD severity is defined according to MAGIC criteria. It will be notified by specifying the location (liver, skin, gut …), the severity score (II to IV), the treatment applied and the efficacy of treatment. GvHD occurrence will be notified every week until D30 (minimum) or until hospital discharge, then monthly until D180 and at D270, D360, D540 and D720.
Cumulative incidence of chronic GvHD | At Day 720 after allogeneic hematopoietic stem cell transplantation
  Chronic GvHD severity will be defined according to NIHCC criteria. It will be notified by specifying the location (liver, skin, gut …), the severity score (II to IV), the treatment applied and the efficacy of treatment. GvHD occurrence will be notified every week until ungraftment, then monthly until D180 and at D270, D360, D540 and D720.
Transplant-Related Mortality | At Day 180, Day 360 and Day 720 after allogeneic hematopoietic stem cell transplantation
  Transplant-related mortality is defined as death due to causes unrelated to the underlying disease.
Cumulative incidence of infections | At Day 360 after allogeneic hematopoietic stem cell transplantation
  Infectious complications will be notified every week up to day 30 (minimum) or until hospital discharge, then every month up to D180 and from D270 to D360, according to the existence of a documented bacteraemia, germ resistance, type and number of days of curative antibiotherapy used; the existence of a documented fungal infection and the type and number of days of curative antifungal treatment; the existence of a documented viral infection and the type and number of days of curative antiviral treatment; the need of an intensive care unit transfer due to an infectious complication.
Severe infections description | From the day of inclusion to Day 360 after allogeneic hematopoietic stem cell transplantation
  Severe infections will be defined according to GREFIG score : bactearemia with severe sepsis, complex bactearemia (with deep organ involvement), candidemia (at least one positive blood culture) with sepsis or deep infected site, proven or probable aspergillosis pneumonia, severe varicella-zoster virus infection (involvement of a deep organ or associated coagulopathy), any viral encephalitis, CMV infection with lung or digestive location, Pneumocystis jiroveci pneumonia, toxoplasmosis with involvement of organ or central nervous system, any acute pneumonia with PaO2 less than or equal to 65mmHg, any sepsis requiring transfer to an intensive care unit.
Impact of Fecal Microbiota Transplantation (FMT) on multi-resistant bacteria, extended-spectrum beta-lactamases and Clostridium difficile infection | At Day 360 after allogeneic hematopoietic stem cell transplantation
  Impact of FMT on multi-resistant bacteria, extended-spectrum beta-lactamases and Clostridium difficile infection will be assessed by evaluation of persistence or disappearance of these pathogenic bacteria after FMT.
Unexpected event description that could be in relation with FMT of Fecal Microbiota Transplantation (FMT) | From the day of FMT to Day 360 after allogeneic hematopoietic stem cell transplantation
  Each unexpected event that could be in relation with FMT will be notified: abdominal pain, diarrhea, bacterial translocation or any adverse effect attributed to the enema.
Quality of life assessment | at Day -7, Day 30, Day 90, Day 180, Day 360 and Day 720 after allogeneic hematopoietic stem cell transplantation
  The quality of life will be auto-evaluated by the patients using a validated questionnaire: European Organisation for Research and Treatment of Cancer- Quality of Life Questionnaire-Core 30 (EORTC-QLQ-C30). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Analysis the intestinal microbiota in patients | Before the conditioning regimen, before the FMT and at Day 30, Day 90 and Day 360 after white blood cells recovery
  The intestinal microbiota composition and diversity will be assessed by 16S-rRNA sequencing performed prospectively in all patients with FMT and without FMT.
Analysis the intestinal microbiota in stool donnors | At the time of the first stool donnation between Day 7 to Day 55 after the inclusion
  The intestinal microbiota composition and diversity will be assessed by 16S-rRNA sequencing performed prospectively in all stool donnors.
Blood collection for a metabolomic study in patients | Before the conditioning regimen, before the FMT and at Day 30, Day 90 and Day 360 after white blood cells recovery
  A blood collection will be set up from blood samples collected on patients from both groups. These samples will be used for a metabolomic study (tryptophan, indoleamine 2,3-dioxygenase, short chain fatty acid, bile acids).
Blood collection for an analysis of anti-microbiota IgG and IgA in patients | Before the conditioning regimen, before the FMT and at Day 30, Day 90 and Day 360 after white blood cells recovery
  A blood collection will be set up from blood samples collected on patients from both groups. These samples will be used for an analysis of anti-microbiota IgG and IgA.
Blood collection for a metabolomic study in stool donnors | At the time of the first stool donnation between Day 7 to Day 55 after the inclusion
  A blood collection will be set up from blood samples collected on stool donnors. These samples will be used for a metabolomic study (tryptophan, indoleamine 2,3-dioxygenase, short chain fatty acid, bile acids).
Blood collection for an analysis of anti-microbiota IgG and IgA in stool donnors | At the time of the first stool donnation between Day 7 to Day 55 after the inclusion
  A blood collection will be set up from blood samples collected on stool donnors. These samples will be used for an analysis of anti-microbiota IgG and IgA.
Stool collection for an analysis of the virome in patients | Before the conditioning regimen, before the FMT and at Day 30, Day 90 and Day 360 after white blood cells recovery
  A stool collection will be carried out from stool samples collected on patients from both groups.These samples will be used for an analysis of the virome evolution.
Stool collection for an analysis of the virome in stool donnors | At the time of the first stool donnation between Day 7 to Day 55 after the inclusion
  A stool collection will be carried out from stool samples collected on stool donnors.These samples will be used for an analysis of the virome evolution.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques-Olivier BAY, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand; Stéphanie NGUYEN, MD, PhD, Principal Investigator — Groupe hospitalier Pitié-Salpêtrière, Paris
Locations (20):
- France (20):
  - Service d'Hématologie Clinique et Thérapie Cellulaire CHU Amiens Picardie - Site Sud, Amiens
  - Service Maladies du sang CHU Angers, Angers
  - Hématologie clinique CHU Besançon, Besançon
  - Plateforme d'Investigation Clinique / Centre d'Investigation Clinique - Inserm 1405, CHU Gabriel Montpied Clermont-Ferrand, Clermont-Ferrand
  - Service de thérapie Cellulaire et d'Hématologie Clinique Adulte CHU Estaing - Clermont-Ferrand, Clermont-Ferrand
  - Service hématologie CHU Grenoble, Grenoble
  - Service des Maladies du sang Hôpital HURIEZ, CHRU de Lille, Lille
  - Service de thérapie cellulaire et l'hématologie clinique adulte CHU Limoges, Limoges
  - Service d'Hématologie Centre Hospitalier Lyon Sud, Lyon
  - Service d'Hématologie et de Médecine interne Hôpital Brabois CHRU Nancy, Nancy
  - Service d'Hématologie Clinique CHU Nantes, Nantes
  - Service d'hématologie clinique, département de greffe de moelle CHU Nice, Nice
  - Service d'Hématologie Adultes Hôpital Necker, Paris
  - Service d'Hématologie clinique Hôpital Pitié-Salpêtrière, Paris
  - Service d'hématologie greffe Hôpital St Louis, Paris
  - Hématologie clinique et thérapie cellulaire Hôpital Haut-Lévèque, Pessac
  - Service d'hématologie greffe Hôpital St Louis, Poitiers
  - Département d'hématologie CAC Rouen, Rouen
  - Hématologie clinique Institut de Cancérologie de la Loire, Saint-Etienne
  - IUC T - Oncopôle, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Full protocol, participant-level data, statistical codes, trial datasets and analyses will be made available on request from the corresponding author after examining the request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study, on request from the corresponding author after examining the request.
Access Criteria: On request from the corresponding author after examining the request.

REFERENCES:
- [Derived] Douge A, Ravinet A, Corriger A, Cabrespine A, Wasiak M, Pereira B, Sokol H, Nguyen S, Bay JO. Faecal microbiota transplantation to prevent complications after allogeneic stem cell transplantation for haematological malignancies: a study protocol for a randomised controlled phase-II trial (the FMT-allo study). BMJ Open. 2023 May 2;13(5):e068480. doi: 10.1136/bmjopen-2022-068480. PMID 37130682